Official Title: Grasping Function After Spinal Cord Injury

ClinicalTrials.gov ID: NCT03447509

ICF document version date: 8/29/2024

| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

#### KEY SUMMARY INFORMATION ABOUT THIS STUDY

You are being invited to take part in a research study that is being funded by the Department of Veterans Affairs. Before you decide to take part, it is important for you to know why the research is being done and what it will involve. This includes any potential risks to you, as well as any potential benefits you might receive. This study involves the use of TMS (transcranial magnetic stimulation) and is not FDA approved for how it is being used in this study.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

By doing this study, we hope to learn how to facilitate recovery of arm and hand movements by using stimulation and exercise training.

Your participation in this research could vary. If you choose to participate in experiment 1 you will be asked to participate in 2-4 sessions lasting 1.5-3 hours each separated by a few days. If you choose experiment 2, you will be asked to complete 20 training sessions each lasting for 2-3 hours. You will be asked to attend 3-5 sessions per week over 6 months.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

This study is being conducted to determine if stimulation and exercise training can enhance the beneficial effects of arm and hand training on improving limb function in persons with spinal injury. We have information suggesting that stimulation and exercise training can improve arm and hand motor function in persons with spinal injury. For a complete description of benefits, refer to the Detailed Information section of this form. Your participation may help medical research determine methods for improving hand movement and function following spinal cord injury. The information obtained from your participation may help others in the future.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

As with any experimental procedure, there may be adverse events that are currently unknown and certain of these unknown risks could be permanent, severe, or life threatening. Procedures in this study may cause all, some or none of the risks or adverse events listed. Rare, unknown, or unforeseeable (unanticipated) risks also may occur. There are no direct benefits to you from your taking part in this research study. However, the information we get from this study might help us treat future patients.

The most common risks of participation are:

- Mild discomfort at the stimulation site and associated muscles
- You may get mildly tired during the evaluations
- Mild headache from the stimulation

Please see "POSSIBLE RISKS OR DISCOMFORTS" below for all risks and discomforts.

Hines ICF Version Date: 8/29/2024

| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

# WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

The person in charge of the study (Principal Investigator) is Monica Perez. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study her contact information is: 312-238-2886 Monica.perez@va.gov

#### DETAILED INFORMATION ABOUT THE STUDY

#### WHAT IS THE PURPOSE OF THIS STUDY?

The study is being conducted to look at recovery of arm and hand movements by using TMS (Transcranial magnetic stimulation), electric stimulation, and exercise training. You are being asked to participate in a research study investigating the effects of stimulation and upper limb training on arm strength and function. We have information suggesting that stimulation and exercise training can improve arm and hand motor function in persons with spinal injury. TMS is a non-invasive procedure that uses a coil placed against your scalp to create magnetic fields to stimulate nerve cells in the brain.

**HOW LONG WILL I BE IN THE STUDY?** This research study is expected to take approximately 2 years. Your individual participation in the project will take anywhere from 2 days to 26 days depending on which experiment you are in. These days can span out across weeks and months if needed.

# WHAT WILL HAPPEN IF I TAKE PART IN THE STUDY?

We anticipate screening at the Hines VA and at the Shirley Ryan Ability Lab leased VA space. We project screening 100 SCI subjects and 75 control subjects. We plan to enroll 12 SCI in experiment 1 and 48 SCI in experiment 2. We plan to enroll 12 control subjects in experiment 1 and 48 control subjects in experiment 2. Not everyone will meet the inclusion criteria.

In experiment 1, you will be asked to participate in 2-4 sessions lasting 1.5-3 hours each in a random order separated by a few days. These sessions will include the following: (1) TMS applied during precision (like pinching a small object), (2) TMS applied during power grip (like making a fist), (3) a startle response applied during precision and (4) a startle response applied during power grip. (5) EMG (electromyography, where an electrode needle or sticker is inserted into the muscle) applied during precision (like pinching a small object) as well as power grip (like making a fist). You will be placed into one of the groups without knowing which group you are in, this is called randomization.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

# Experiment 1 (Crossover design)



# In Experiment 1 the following procedures will be conducted:

- TMS stimulation on your scalp
- Recording of your muscle activity
- Your startle response to loud noises
- Electrical stimulation on your wrist
- An assessment of your hand function
- A sensory test

# For SCI participants only:

 An exam to determine your abilities to move your muscles and to test your feeling using a clinical exam, ASIA.

These measurements are described in detail below in "Study Procedures".

In experiment 2, you will be asked to complete 20 training sessions each lasting for 2-3 hours. You will be asked to attend 3-5 sessions per week. Additional sessions may be needed if sessions are missed or not completed. You will be randomly placed into one of the four study groups. In these sessions you will not know when you are receiving real stimulation or sham (fake) stimulation. There is a 50% chance (like flipping a coin) of receiving fake stimulation. For the exercise training you will be asked to complete different arm and hand movements. You will be asked to complete 2 testing sessions before the 20 training sessions and 2 testing sessions after the training sessions.

### Experiment 2 (Controlled design)



For SCI participants only:

 An exam to determine your abilities to move your muscles and to test your feeling using a clinical exam, ASIA.

 You will be asked to complete 2 surveys (1) Self-care subscale of the Spinal Cord Independence Measure-Version III (SCIM) and (2) The Capabilities of Upper Extremity (CUE).

# In Experiment 2 the following procedures will be conducted:

- TMS stimulation on your scalp
- Recording of your muscle activity
- Your startle response to loud noises
- Electrical stimulation on your wrist
- An assessment of your hand function
- A sensory test
- Arm and hand exercise training


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

#### STUDY PROCEDURES

If you are interested in participating, we will first review our eligibility criteria with you, the informed consent, complete an intake questionnaire including past medical and surgical history.

**Screening Procedures:** During the in-person screening session, which may last up to 1 hour, you may be asked to complete some or all of the following procedures:

- · Sign the informed consent document before any procedures are performed
- A general screening and medical intake questionnaire
- · A strength assessment of your arms, and hands
- A variety of hand positions (making a cylinder, lateral key pinch or tip to tip pinch)
- Sensation testing of your upper body
- Testing to determine your response to TMS
- A questionnaire to evaluate if your injury is complete or incomplete (SCI only)

We will encourage you to ask any questions you may have during this time.

To evaluate your responsiveness to TMS, we will deliver a few stimulations to your brain and record the response from the muscle being tested. This is done to see if we can get specific recordings from different muscles. During this testing you might feel movement or a twitch in your muscles.

#### **Experimental Procedures for all participants:**

If you qualify to take part in this research study, you will be asked to participate in experiment 1, experiment 2, or both. These experiments will take place at the Hines Spinal Cord Building (building 128), room A150. The research staff will work with you to schedule times when you are available. You may also be tested in lab space at Shirley Ryan Ability Lab located at 355 E Erie St, Chicago, IL 60611.

Depending on the experiment and group combination that you are assigned to, you may be asked to complete any of the below tasks:

**Electromyography (EMG):** Recording electrodes will be attached to either the surface of your skin over selected muscles or to the muscle directly using sterile needles, to record the activity within these muscles. Customized equipment will be attached to your arms and fingers to measure your strength and ability to move.

**Transcranial Magnetic Stimulation (TMS):** A wire coil will be placed over your head. When activated, this coil will generate a magnetic pulse over a specified area of your head. You may also feel a small twitch of the muscles in your arm, face or your hand. Several series of pulses will occur over the course of the session.

**Peripheral Nerve Stimulation (PNS):** Peripheral nerve stimulation will involve placing a small device on the surface of your skin that will deliver pulses of electricity on the limbs. These pulses may feel strange, but should not feel uncomfortable.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

Cervicomedullary Motor Evoked Potentials (CMEPs): We will deliver pulses of electrical stimulation near the mastoid process, which is the bone behind the ear. These pulses may feel strange, but should not feel uncomfortable.

**Electrical Perceptual Threshold (EPT):** EPT is a sensory exam that uses small electrical pulses to examine your ability to feel the stimulation.

Chedoke Arm and Hand Activity Inventory (CAHAI): We will examine the ability of your hand and harm to perform certain tasks.

**Jebsen Taylor Hand Function Test (JTT):** We will examine your hand function by using simulated activities of daily living.

Pinch Grip Strength (Force): We will assess the strength you can produce with your arm and hand

Hand Assessments: Periodically during testing, we will evaluate your ability to use your arms and hands. You will be asked to complete a series of tasks such as stacking checkers, turning over cards, squeeze a device to determine how strong your grip is, and see how well you are able to feel sensations on the surface of your skin.

# For SCI participants:

**ISNCSCI Exam (ASIA):** You will be asked to complete an ASIA exam which evaluates your muscle and sensory function by looking at different points along the body. It checks to see if you can sense light touch, and if you can tell the difference between sharp and dull sensation.

**Surveys:** The following two questionnaires will be given to you before your first training session and then again after your last training session. You do not have to answer any questions you do not want to. They will each take approximately 5 minutes to complete:

- (a) Self-care subscale of the Spinal Cord Independence Measure- Version III (SCIM). In this questionnaire we will ask you about your ability to complete basic daily functions using your upper such as feed, bathe upper body, dress upper body, and groom.
- (b) The Capabilities of Upper Extremity (CUE).

In this questionnaire, we will ask you about your ability to perceive how much function you have with your hands and arms by your ability to reach or lift, pull and push with arms, moving and positioning arm and wrist, and the ability to use hands and fingers.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

#### WHAT IS EXPECTED OF ME IF I TAKE PART IN THIS STUDY?

- Keep your study appointments.
- If you miss an appointment, please contact the investigator or research staff to reschedule as soon as you know you will miss the appointment.
  - Tell the investigator or research staff if you believe you might be pregnant or might have gotten your partner pregnant.
  - Complete your diaries as instructed.
  - Complete your questionnaires as instructed.
  - Ask questions as you think of them.
  - o While participating in this research study, do not take part in any other research project without approval from the investigators. This is to protect you from possible injury from things such as extra blood drawing, extra X-rays, or potential drug interactions. Taking part in other research studies without first discussing it with the investigators of this study may invalidate the results of this study, as well as that of the other studies.

We may request copies of medical records from outside non-VA facilities. A VA Form Letter 10-212 will need to be signed for each different non-VA entity from which records will be requested.

### WHAT POSSIBLE RISKS OR DISCOMFORTS MIGHT I HAVE IF I TAKE PART IN THIS STUDY?

Any procedure has possible risks and discomforts. The procedures in this study may cause all, some, or none of the risks or side effects listed. Rare, unknown, or unexpected risks also may occur. There is always a chance that any procedure can harm you. Risks of the usual care you receive are not risks of this study. Those risks are not included in this consent form. You should talk with your health care providers if you have any questions about the risks of usual care.

# For Women of Child-bearing Potential:

Magnetic fields reduce rapidly with distance, and it is unlikely that a fetus might be affected by the use of TMS. However, the effects of TMS during pregnancy are unknown. For this reason, pregnant women are excluded from this study. There may be unforeseeable (unanticipated) risks to the participant (or to the unborn child) if the participant is pregnant or becomes pregnant during the study.

Prior to performing TMS procedures in each session, female participants will be asked about their pregnancy status, and they will be informed that the effects of TMS during pregnancy are unknown. Participants who are uncertain about their pregnancy status and want to participate in the study will receive a urine pregnancy test prior to undergoing any TMS procedures. For these individuals, at each research visit, we will document pregnancy status and offer a urine pregnancy test if warranted. Acceptable forms of birth control are:

- Complete abstinence (not having sexual intercourse with anyone)
- An oral contraceptive (birth control pills)
- Norplant

IRBnet# 1517521


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| | Page 7 of <b>13</b> |
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

Depo-Provera

- · A condom with spermicide
- A cervical cap with spermicide

# Risks of Muscle Activity Recording (EMG):

Mild discomfort, such as a mild itching sensation may be felt under the electrodes that register the response in your muscles. The possibility of this is infrequent (occurring in 1-10%, or 1-10 out of 100 people). We will clean the area with alcohol and use standard, hospital grade electrodes.

#### Risks of Intramuscular Needle EMG:

The major risks for intramuscular needle EMG recording are infrequent (1-10%) but may include minor pain, mild bleeding and infection. The risk of infection will be minimized by using sterilized needles

# Risks of Transcranial Magnetic Stimulation (TMS):

There is the rare possibility (occurs in less than 1%, or less than 1 out of 100 people) that TMS could cause a seizure. When assessing your eligibility to participate in this research, we ask specific questions that help us to determine whether or not you would be more likely to experience this particular risk. Individuals who are at increased risk for this complication will be excluded.

Additional, infrequent risks (< 2%) associated with TMS include mild headache, mild discomfort at the stimulation site and associated muscles, weakness, tingling, and a feeling of tiredness.

The stimulation produces a clicking sound. To reduce any discomfort due to the volume of this sound, you will be required to use earplugs or earphones to protect hearing acuity.

During TMS testing the coil may get warm. It may feel about the same as a heating pad on low or medium setting. This may be uncomfortable but should not be painful. The frequency of this event depends of the stimulation intensity and number of pulses tested.

In the unlikely event of a seizure, the rapid response team or 911 will be called.

# Risks of the Peripheral Nerve Stimulation and Recording:

Mild discomfort, such as an itching sensation may be felt under the electrode that stimulates your wrist or under the electrodes that register the response in your muscles. The possibility of this is infrequent (occurring in 1-10%, or 1-10 out of 100 people). We will clean the area with alcohol and use standard, hospital grade electrodes. Another risk of the nerve stimulation used in this research is that you might feel mild pain, if pain fibers could be activated.

# Risks of the Physical Assessments:

It is possible that you may get mildly tired during the evaluations. To minimize the risk, you will have resting periods as needed.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| | Page <b>8</b> of <b>13</b> |
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

#### Risks of CMEPs:

Mild discomfort, such as an itching sensation may be felt under the electrode that stimulates your wrist or under the electrodes that register the response in your muscles. The possibility of this is infrequent (occurring in 1-10%, or 1-10 out of 100 people). A higher stimulus intensities will be used near the bone behind the ear (mastoid process) to create a motor response in the muscles of the upper and lower limbs. This might result in some discomfort for some participants. In order to keep the discomfort at a minimum, stimulation will start at a very low intensity and increase slowly.

**Startle:** Loud noises and visual stimuli can precipitate PTSD. If you feel this procedure has affected your PTSD, please contact your mental health provider.

In the event of an emergency 911 or the hospital rapid response team will be called to provide assistance.

#### WHAT ARE THE POSSIBLE BENEFITS OF THIS STUDY?

There are no direct/personal benefits to you from your taking part in this research study. However, the information we get from this study might help us treat future patients.

# WHAT OTHER CHOICES DO I HAVE IF I DO NOT WANT TO JOIN THIS STUDY?

Taking part in this study is completely voluntary. You may choose not to take part in this study or leave this study at any time. This is not a treatment study. Your alternative is not to participate in this study. This will not affect your care or benefits at Hines VA. Your decision will not have any impact on your participation in other studies and will not result in any penalty or loss of benefits to which you are otherwise entitled.

You can leave the research at anytime and it will not be held against you. You may withdraw, at any time, your consent for participation in this research study. Any identifiable research or medical information recorded for, or resulting from, your participation in this research study prior to the date that you formally withdrew your consent may continue to be used and disclosed by the investigators for the purposes described above.

#### CONFIDENTIALITY

HOW WILL MY PRIVATE INFORMATION BE PROTECTED?

This research study involves the recording of current identifiable medical information. The information that will be recorded will be limited to information concerning the purpose of this research and your safety. All records related to your involvement in this research study will be stored in a locked file cabinet.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

Your identity on these records will be indicated by a case number rather than by your name, and the information linking these case numbers with your identity will be kept separate from the research records.

As with any research, there is always a minor risk of a breach of confidentiality. That is, in very rare cases, people not associated with this research study may, inadvertently, see your identifiable research results. We will do everything in our power to prevent this from happening by keeping all research records in locked files. Identifiable electronic information related to your participation will be stored on restricted access password protected servers.

There are times when we might have to show your records to other people. For example, someone from the Office of Human Research Protections (OHRP), the Government Accountability Office, the Office of the Inspector General, the VA Office of Research Oversight, VA Office of Research and Development, the VA Institutional Review Board (IRB), our local Research and Development Committee, authorized members of the Human Research Protection Program, and study monitors may look at or copy portions of records that identify you.

In unusual cases, the investigators may be required to release identifiable information (which may include your identifiable medical information) related to your participation in this research study in response to an order from a court of law.

You will not be identified by name in any publication of the research results unless you, a POA, or a LAR sign a separate consent form giving permission (release).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. The clinical trial number, NCT03447509, can be used to allow for the study to be easily looked up. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. The study is listed as B2474-R, Grasping Function after Spinal Cord Injury.

#### Health Information Portability and Accountability Act (HIPAA)

There are rules to protect your private information. Federal and state laws and the federal medical Privacy Rule also protect your privacy. By signing this form, you provide your permission called your 'authorization,' for the use and disclosure of information protected by the Privacy Rule. If you require a POA for participation in this study, a separate VA HIPAA Authorization form 10-0439, will need to be signed.

The research team working on the study will collect information about you. This includes things learned from the procedures described in this consent form. The study team may also collect other information including your name, address, date of birth, and information from your medical records such as HIV status, drug, alcohol or STD treatment, genetic test results or mental health treatment.


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

The research team may also need to disclose the information to others as part of the study progress. Others may include the following: the Office of Human Research Protections, the Government Accountability Office, the Office of the Inspector General, the VA Office of Research Oversight, VA Office of Research and Development (sponsor), the VA Institutional Review Board (IRB), the US Food & Drug Administration (FDA), study monitors, authorized representatives of the Hines VA Research Administration and Hines Human Research Protections Program.

Your health information disclosed pursuant to this authorization may no longer be protected by Federal laws or regulations and may be subject to re-disclosure by the recipient.

While this study is being conducted you will not have access to your research related health records.

This will not affect your VA healthcare, including your doctor's ability to see your records as part of your normal care and will not affect your right to have access to the research records after the study is completed.

You can revoke this authorization, in writing, at any time. To revoke your authorization, you must write to the Release of Information Office at Hines VA or you can ask a member of the research team to give you a form to revoke the authorization. Your request will be valid when the Release of Information Office receives it. If you revoke this authorization, you will not be able to continue to participate in the study. This will not affect your rights as a VHA patient to treatment or benefit outside of the study.

If you revoke this authorization, The Investigator, Monica Perez, PhD, and her research team can continue to use information about you that was collected before receipt of the revocation. The research team will not collect information about you after you revoke the authorization.

Treatment, payment or enrollment/eligibility for benefits cannot be conditioned on you signing this authorization. This authorization will expire at the end of the research study unless revoked prior to that time.

### COSTS TO PARTICIPANTS AND PAYMENT

There is no cost to you for your participation in this research study.

You will not be charged for any treatments or procedures that are part of this study. If you usually pay co-payments for VA care and medications, you will still pay these co-payments for VA care and medications that are not part of this study.

Payment Offered for Participation If you agree to take part in this research study, you will be paid \$10 per hour. All payments will be made by direct deposit via Electronic Funds Transfer (EFT). The EFT process will use your social security number. Veterans who are unable to utilize this option (i.e., do not


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

have a bank account or the ability to get a Direct Express Debit card) may not be able to receive compensation. You will have an opportunity to discuss these options before you consent to participate in the study.

#### WHAT WILL HAPPEN IF I AM INJURED BECAUSE OF MY BEING IN THE STUDY?

If you are injured as a result of taking part in this study, the VA will provide necessary medical treatment at no cost to you or your insurance unless the injury is due to non-compliance by a study participant with study procedures or if the research is conducted for VA under contract with an individual or non-VA institution. If you have additional questions, please contact the Study Investigator, or contact Hines VA and ask for the ACOS/Research.

You do not give up any of your legal rights and you do not release the VA from any liability by signing this form.

If you should have a medical concern or get hurt or sick as a result of taking part in this study, call:

DURING THE DAY:

| | at | and |
|--------------|----|-----|
| AFTER HOURS: | | |
| | at | |

#### DO I HAVE TO TAKE PART IN THE STUDY?

Taking part in this study is completely voluntary. You may choose not to take part in this study or leave this study at any time. This is not a treatment study. Your alternative is not to participate in this study. This will not affect your care or benefits at The Hines VA. Your decision will not have any impact on your participation in other studies and will not result in any penalty or loss of benefits to which you are otherwise entitled.

### RIGHT OF INVESTIGATOR TO TERMINATE PARTICIPATION

The researcher may remove you from the study if she believes that staying in the study is no longer in your best interest. If you stop being in the study, the study staff and the study doctor will stop collecting your health information. Although they will stop collecting new information about you, they may need to use the information they have already collected to evaluate the study results. If you start the study and then you cancel your permission, you will not be able to continue to participate in the study. We will tell


| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

you about any new information or changes in the study that might change your decision to stay in the study. You may be asked to sign a new consent form if this occurs.

# **FUTURE USE OF DATA OR SPECIMEN**

The data collected as part of this research study, even if identifiers are removed, will not be used or distributed for future research studies.

#### WHO DO I CONTACT ABOUT THIS STUDY IF I HAVE QUESTIONS?

If you have questions about your rights as a study participant, or you want to make sure this is a valid VA study, you may contact the Edward Hines Jr. VA Hospital IRB Office 708-202-2811. This is the Board that is responsible for overseeing the safety of human participants in this study. You may call the Edward Hines Jr. VA Hospital IRB Office if you have questions, complaints or concerns about the study or if you would like to obtain information or offer input.

has explained

#### AGREEMENT TO PARTICIPATE IN THE RESEARCH STUDY

| the research study to you. You have been told of the risks or discomforts and possible benefits of the study. You have been told of other choices of treatment available to you. You have been given the chance to ask questions and obtain answers. | | | |
|---|---|---|---|
| | By signing this document below, you voluntarily consent to participate in this study and authorize the use and disclosure of your health information in the study. You also confirm that you have read this consent or it has been read to you. You will receive a copy of this consent after you sign it. | | |
| I agree to participate in this research study as has been explained in this form. | | | |
| | Participant's Name | Participant's Signature | <br>Date |
| | Name of Person Obtaining | Signature of Person Obtaining | |
| | consent | Consent | Date |


IRBnet# 1517521

Dr./Mr./Ms

| Department of Veterans Affairs | Edward Hines Jr Combined Informed<br>Consent Form and HIPAA Authorization<br>Template<br>Version Date: 8/29/2024 |
|---|---|
| Participant Name: | Date: |
| Title of Study: Grasping Function after Spinal Cord Injury | |
| Principal Investigator: | |

| I agree to participate in this research study as has been explained in this form. | | |
|---|---|---|
| Participant's Name | Participant's Signature | Date (coordinator initial) |
| Witness #1 Name | Witness #1 Signature | <br>Date |
| Witness #2 Name | Witness #2 Signature | <br>Date |
| Name of Person Obtaining consent | Signature of Person Obtaining Consent | Date |
